CLINICAL TRIAL: NCT00897611
Title: Identification of Hypermethylated Serum Tumor DNA in High Grade Glioma Patients and Correlation With Magnetic Resonance Imaging Findings
Brief Title: Tumor DNA and MRI/CT Scan Findings in Patients With Grade III or Grade IV Malignant Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); North American Brain Tumor Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NABTT-0402 CDR0000462562; U01CA062475 (NIH); NABTT-0402
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: High Grade Glioma
Keywords: adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; recurrent adult brain tumor; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — DNA Methylation; Blood Specimen Collection; Polymerase Chain Reaction; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: DNA methylation analysis
  Other Names: blood collection
Procedure: polymerase chain reaction
  Other Names: blood collection
Procedure: computed tomography
  Other Names: CT scan
Procedure: magnetic resonance imaging
  Other Names: MRI scan

SUMMARY:
RATIONALE: Studying levels of tumor DNA in the samples of blood from patients with cancer may help doctors find out whether the cancer has grown and how much.

PURPOSE: This laboratory study is comparing levels of tumor DNA with MRI and CT scan findings to measure cancer growth in patients with grade III or grade IV malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate changes in the level of serum tumor-specific DNA over time with changes in brain tumor size as measured by serial MRI or CT scans in patients with grade III-IV malignant gliomas.

OUTLINE: This is a multicenter study.

Blood samples are collected from patients at baseline and every 2 months thereafter. Tumor and nontumor plasma is extracted. Plasma samples are analyzed by polymerase chain reaction (PCR) to assess the p16_ink4a, p73, and O ^6-MGMT gene promoter methylation profile. Quantitative realtime PCR is performed on samples with tumor-specific DNA to determine the plasma concentrations of each methylated tumor-specific gene and the total plasma tumor-specific DNA concentration. Patients also undergo MRI or CT scans every 2 months.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant brain tumor

  * One of the following grade III or IV supratentorial gliomas:

    * Anaplastic astrocytoma
    * Anaplastic oligodendroglioma
    * Glioblastoma multiforme
* Newly diagnosed or recurrent disease
* Planning to undergo anticancer therapy on a New Approaches to Brain Tumor Therapy (NABTT) Consortium clinical trial

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-04; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Total plasma glioma-specific DNA concentration | every 2 months until death
Tumor size | every 2 months until death

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Kyle Weaver, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center